CLINICAL TRIAL: NCT05847140
Title: A Non-interventional Multi-country Cohort Study to Assess the Safety of EVUSHELD™ (Tixagevimab/Cilgavimab) During Pregnancy
Brief Title: A Non-interventional Multi-country Cohort Study to Assess the Safety of EVUSHELD™ During Pregnancy
Acronym: O-STEREO
Status: Withdrawn | Type: Observational
Why Stopped: The MAH's proposal to remove the Study from the RMP is based on the change in circulating COVID-19 variants, which has led to a suspension of EUA and significant decrease in the use of EVUSHELD.
Sponsor: AstraZeneca (Industry)
Collaborators: Aetion, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: D8850R00006
Record Dates: First submitted 2023-02-21; First posted 2023-05-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy; Pregnant Women; Pregnancy Outcome
Keywords: Pregnancy outcome; evusheld; pregnancy exposure; immunocompromised condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Evusheld exposed pregnancies: A pregnancy is considered exposed to EVUSHELD if 1 of 2 conditions are met: (1) EVUSHELD was received during the 36-week period [reflective of roughly 3 half-lives of EVUSHELD] prior to LMP, or (2) EVUSHELD was received on/after LMP during the exposure ascertainment period, which will vary based on the outcome of interest.

SUMMARY:
Multi-country, non-interventional cohort study.The objective of the study is to characterise the risk of pregnancy and offspring (neonatal and infant) outcomes in pregnancies with and without exposure to EVUSHELD (used as a treatment or prophylaxis) among women of child-bearing indicated for such treatment in the real-world setting, using secondary data from US, France and Canada.

DETAILED DESCRIPTION:
This is a multi-country, non-interventional cohort study in pregnancies exposed to EVUSHELD and pregnancies unexposed to EVUSHELD among women eligible for EVUSHELD. The study will be conducted within secondary data sources (administrative claims, electronic medical records (EMR) and/or registry data). For each country, the overall study period will span 12 months prior to the country-specific EVUSHELD availability until the end of the data cut or 31 March 2027, whichever is earlier.

The study will include pregnancies in individuals eligible for EVUSHELD therapy in each country in the selected datasets, including pregnant individuals aged 18 to 49 years with a high-risk condition documented in the 12 months prior to the start of the pregnancy, defined as the first day of the last menstrual period (LMP).

ELIGIBILITY:
Inclusion Criteria:

* Female sex at LMP
* Age 18-49 years at LMP
* Continuous coverage/clinical activity (dependent on data source type) within the confounder ascertainment period
* LMP date falls within the LMP eligibility period
* Occurrence of at least one of the following high-risk conditions during the confounder ascertainment period
* Immunocompromised conditions:

  * Cancer (active solid cancer, blood cancer, or receipt of chemotherapy, immunotherapy, or radiotherapy)
  * Solid organ transplant
  * HIV/AIDS
  * Prolonged systemic corticosteroid use (15-20 mg of prednisone equivalents for greater than 2 weeks)
  * Receipt of T or B cell depleting therapy, anti-Tumour Necrosis Factor (anti- TNF), or other immunosuppressive agents
  * Receipt of stem cell transplant
  * Receipt of gene cell therapy of the CAR-T cell type
  * Congenital immunodeficiency, primary immune deficiencies (treatment with subcutaneous or intravenous immunoglobulins - and/or immunodeficiency diagnosis codes), severe or combined immunodeficiency (including transplanted
  * Severe combined immunodeficiency [SCID] where immunoglobulin replacement is required)
  * Other autoimmune conditions and immune-mediated inflammatory disorders (such as systemic lupus erythematosus, Crohn's disease, ulcerative colitis).
* Conditions that increase risk of COVID-19 disease progression

  * Severe risk of COVID-19 disease progression: sickle cell disease, chronic lung disease (ie, chronic bronchitis, Chronic obstructive pulmonary disease [COPD], cystic fibrosis, emphysema with dyspnoea on exertion), chronic kidney disease, cardiovascular diseases (ie, heart failure, coronary artery disease, cardiomyopathies), moderate to severe asthma, Down syndrome, rare neurological conditions (ie, multiple sclerosis, motor neurone disease, myasthenia gravis, Huntington's disease), gestational diabetes requiring medication
  * Moderate risk of COVID-19 disease progression: type I or II diabetes, obesity, chronic liver disease, congenital heart disease

Exclusion Criteria:

* Multifoetal pregnancies are defined by the presence of any International Classification of Diseases (ICD-10) diagnosis code, any position indicating presence of more than one foetus (see code list) on the hospital record throughout the pregnancy episode
* Use of in vitro fertilisation or other assisted reproductive technology in the 36 weeks prior LMP as identified by ICD-10 diagnosis code "pregnancy resulting from assisted reproductive technology" or related procedure codes indicating in vitro fertilisation (IVF) or assisted reproductive technology (ART) (see code list) on the electronic health records (EHR) or hospital claims records 36 weeks prior to LMP

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: The study will include pregnancies in individuals eligible for EVUSHELD administration in each country, including pregnant females aged 18-49 years with a high-risk condition. Exposed and unexposed pregnancies will be identified from this population for outcome-specific analyses.
  EVUSHELD indication varies from one country to another and may evolve over the course of the study. In order to have a homogeneous study population and maximise its size, all countryspecific EVUSHELD eligibility criteria at the time of protocol development were considered to define the study population.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-27 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Risk of pregnancy outcomes potentially associated with exposure in early pregnancy and measured prior to 20 weeks gestation | Index date to < 20 weeks of gestation
  Spontaneous abortion, Ectopic pregnancy
Risk of pregnancy outcomes potentially associated with exposure anytime during pregnancy and measured anytime during pregnancy | Index date to end of pregnancy (Note: Maternal death outcome ascertainment period is up to 42 days after the end of pregnancy episode (EPE).)
  Maternal Death
Risk of pregnancy outcomes potentially associated with exposure anytime during pregnancy and measured after 20 weeks gestation | Index date to end of pregnancy Note: For preterm birth, the outcome ascertainment period is 20 to 37 weeks of gestation
  Preterm live birth, Stillbirth, Gestational hypertension, Pre-eclampsia, Gestational diabetes
Risk of outcomes in neonates potentially associated with exposure anytime during pregnancy and measured 28 days after birth | Diagnosed within 28 days of birth
  Low birth weight, Small for gestational age, Respiratory distress syndrome in the newborn, Neonatal death
Risk of outcomes in infants potentially associated with exposure anytime during pregnancy and measured within 12 months after birth | From birth to time of death or 12 months of age
  Major congenital malformations, Infant death, Failure to thrive

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home